CLINICAL TRIAL: NCT00508248
Title: Use of Omega 3 Polyunsaturated Fatty Acids Supplements to Maintain Sinus Rhythm in Persistent Atrial Fibrillation
Brief Title: Omega 3 Fatty Acids and Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, AChoy, Senior Clinical Lecturer and Honorary Consultant Cardiologist, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 270605ver3
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Fibrillation
Keywords: omega 3fatty acids
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator): 1 g omega 3 fatty acid supplements
  Interventions: Dietary Supplement: omega 3 fatty acids
- A2 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: omega 3 fatty acids — 1g daily
  Other Names: Omacor
  Arms: A1
Dietary Supplement: placebo — olive oil capsule
  Arms: A2

SUMMARY:
Unlike for ventricular arrhythmias, the role of n-3 PUFAs in atrial arrhythmias has not been fully investigated. A recently published epidemiological study reported that in elderly patients, consumption of fish was associated with a lower incidence of atrial fibrillation over the 12 years of follow-up. This observation may be an indirect effect due to the overall beneficial effort of fish consumption on reducing ischaemic heart disease, however this association persisted after adjustment for confounding characteristics. Clinical data regarding the direct impact of n-3 PUFAs on atrial arrhythmias such as atrial fibrillation/flutter (AF) is lacking. However, as both INa and ICa-L are also in atrial myocytes, similar anti-fibrillatory actions by n-3PUFAs would be expected in atrial fibrillation and we would like to investigate this further. The primary aim of this study is to investigate whether dietary supplements of n-3 PUFA concentrates (1g fish oil/day comprising eicosapentaenoic acid, EPA 46% and docosahexaenoic, DHA 38%)) helps maintain sinus rhythm after cardioversion to normal sinus rhythm in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
The patients. Randomisation. Patients with persistent AF will be recruited from clinic attendees and in-patient hospital patients at Ninewells Hospital and Medical School. A total of 150 patients with AF of more than 7 days duration and scheduled for elective direct current cardioversion will be recruited. The patients will be randomised to receive fish oil supplements (3g/day) or placebo on recruitment for a period of 4 weeks prior to cardioversion and continued after cardioversion until recurrence of AF or until the end of 6 months. All patients will be anticoagulated routinely. Patients on anti-arrhythmic drugs, left atrial size >6 cm, significant mitral valve disease, myocardial infarction in the last 3 months, unstable angina, NYHA IV heart failure, cardiac surgery in the previous 3 months, acute reversible conditions, significant thyroid, hepatic, pulmonary disease, pregnancy or child bearing potential will be excluded from the study.

3.2. End Points of the Study. The primary endpoint will be time to first electrocardiographically confirmed recurrence of atrial fibrillation/flutter lasting more than 10 minutes. Secondary endpoints will be shock number and energy requirements to achieve electrical cardioversion. All patients will give informed consent and approval will be obtained from the Ethics Committee of Ninewells Hospital and Medical School.

3.3. Free n-3 PUFA plasma concentrations On the day of cardioversion, 3mls of venous blood will be obtained for measurement of free n-3 PUFA plasma concentrations.

3.4. Elective Direct current cardioversion and Follow-up Patients will be routinely scheduled for cardioversion (2 per week) as outpatients. Cardioversion will be under conscious sedation (titrated doses of intravenous midazolam) as is the current routine practice in the Department of Cardiology, Ninewells Hospital. Follow-up (with ECG) of cardioverted patients will be weekly in the first month; then 2,3,4,5 and 6 months; and at any time the patients complains of palpitations or other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation
* Post cardioversion

Exclusion Criteria:

* Patients on anti-arrhythmic drugs
* Left atrial size > 6 cm
* Significant mitral valve disease
* Myocardial infarction in the last 3 months
* Unstable angina
* NYHA IV heart failure
* Cardiac surgery in the previous 3 months
* Acute reversible conditions
* Significant thyroid, hepatic, pulmonary disease
* Pregnancy or child bearing potential

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
recurrence of atrial fibrillation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, MD, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital and medical School, Dundee, United Kingdom